CLINICAL TRIAL: NCT06489665
Title: Imaging Quality and Potential Clinical Relevance of Phase Contrast
Brief Title: Imaging Quality and Potential Clinical Relevance of Phase Contrast Mammography In-vivo: a Single-center, Prospective Study
Status: Recruiting | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: Center for Proton Therapy, Paul Scherrer Institute, Villigen,Switzerland (Other); GratXray AG (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2021-00200
Record Dates: First submitted 2024-06-28; First posted 2024-07-08 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer; Microcalcification; Image
Keywords: Mammography
MeSH Terms: conditions — Breast Neoplasms; Calcinosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Mammography finding: Describes the mammography finding in patients prior breast surgery
  Interventions: Diagnostic Test: Experimental Intervention
- Bellona: Describes the finding in the breast tissue samples
  Interventions: Diagnostic Test: Experimental Intervention

INTERVENTIONS:
Diagnostic Test: Experimental Intervention — Mammography in the radiology department is commonly performed using General Electrics Medical Systems Senographe Essential device
  Other Names: control intervention

SUMMARY:
Conventional mammography, breast sonography and breast MRI have specific weaknesses. In particular, mammography has a low sensitivity for the detection of mammary carcinoma in patients with a dense breast. Phase contrast mammography could help to overcome some of these limitations. Observational study.

DETAILED DESCRIPTION:
Category C2 Medicine product without CE label.

Objective(s):

Phase 0: Imaging of mastectomy and breast biopsy samples to validate the image quality and radiation dose. Phase 1: Determination of accurate radiation dose in vivo; dose exposure should remain within the range specified in the investigational brochure. Evaluation of cohort size for phase 2. Phase 2: Assessment of the diagnostic performance of phase contrast mammography compared to conventional digital mammography.

Ouctomes: Sensitivity and specificity of phase contrast mammography compared to conventional digital mammography.

Measurements and procedures:

Phase 0: Phase contrast mammography of the mastectomy, tumorectomy or breast biopsy samples is performed after breast surgery in addition to the standard clinical procedures Phase 1: Phase contrast mammography is performed before the operation in case of known breast carcinoma in addition to the standard clinical procedures Phase 2: Phase contrast mammography is performed directly in the clinical routine. The result is compared with the result of the conventional digital mammography and the ultrasound examination.

Number of Participants with Rationale:

Phase 0: expected to be 30 Phase 1: expected to be 20 Phase 2: expected to be 300 (correct number will be defined according to Phase 1)

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria -Phase 0:

  * >18 years
  * Mastectomy, tumorectomy or biopsy planned
  * Informed consent of the patient

Inclusion criteria -Phase 1:

* >18 years
* BI-RADS 5 (highly suggestive of malignancy at ultrasound or mammography) or 6 (known biopsy proven malignancy);
* Scheduled for mastectomy or breast conserving surgery with radiotherapy.
* Informed consent of the patient

Inclusion criteria - Phase 2:

* >40 years
* undergoing mammography for screening or diagnostic purpose.
* Informed consent of the patient

Exclusion Criteria:

* Exclusion criteria for all three Phases:

  * Breast implants. The women will be asked, if they have a breast-implant.
  * Inability to understand the study procedure due to cognitive or linguistic deficits.

Exclusion criteria for patients, participating in Phase 1 and Phase 2:

* Pregnancy
* Breast-feeding.
* Re-staging after neoadjuvant chemotherapy. Patients who participated in prior research projects with ionizing radiation in the past 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who are scheduled to have a mastectomy, tumorectomy or biopsy
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2024-10-17 (Actual); Primary Completion 2029-09-01 (Estimated); Study Completion 2030-09-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of PCM compared to FFDM represent the primary outcome since the limited sensitivity of mammography, in particular in patients with dense breasts, represents the major limitation of the currently applied FFDM. | 30 month
  The standard reference will be the histologic specimen after biopsy

SECONDARY OUTCOMES:
Lesion extent will be estimated using both PCM and FFDM. Pathological measurements obtained from the surgical specimen will be used as standard of reference. | 30 month
  The aim is to evaluate if PCM, due to the expected improved visibility of the lesions, can allow for a better estimation of lesion extent with subsequent benefit on the preoperative planning.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Frau, Prof, Principal Investigator — University Hospital Zurich, DIR
Locations (2):
- Switzerland (2):
  - University Hospital Zurich - Diagnostic Radiology, Zurich, Canton of Zurich
  - University of Zurich, Zurich

IPD SHARING:
Plan to Share IPD: No